CLINICAL TRIAL: NCT05923424
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of REGN17092, an Anti-SARS-CoV-2 (COVID-19) Monoclonal Antibody, in Adult Healthy Volunteers
Brief Title: A Trial to Learn if Different Doses of REGN17092 Are Safe in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R17092-HV-2312; 2023- 505041-52-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers
Keywords: Severe acute respiratory syndrome coronavirus (SARS-CoV-19); Coronavirus disease 2019 (COVID-19) vaccinated; Omicron variant
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (10):
- Cohort 1 Mid IV Dose (Experimental): Randomized 6:2 for single ascending dose
  Interventions: Drug: REGN17092; Drug: Matching Placebo
- Cohort 3 High IV Dose (Experimental): Randomized 6:2 for single ascending dose
  Interventions: Drug: REGN17092; Drug: Matching Placebo
- Cohort 5 Higher IV Dose (Experimental): Randomized 6:2 for single ascending dose
  Interventions: Drug: REGN17092; Drug: Matching Placebo
- Cohort 6 Low IV Dose (Experimental): Randomized 6:2 for single ascending dose
  Interventions: Drug: REGN17092; Drug: Matching Placebo
- Cohort 2 Mid SC Dose (Experimental): Randomized 6:2 for single ascending dose
  Interventions: Drug: REGN17092; Drug: Matching Placebo
- Cohort 4 High SC Dose (Experimental): Randomized 6:2 for single ascending dose
  Interventions: Drug: REGN17092; Drug: Matching Placebo
- Cohort 7 Low SC Dose (Experimental): Randomized 6:2 for single ascending dose
  Interventions: Drug: REGN17092; Drug: Matching Placebo
- Expansion Cohort 1 (Experimental): Randomized 3:1 for single ascending dose
  Interventions: Drug: REGN17092; Drug: Matching Placebo
- Expansion Cohort 2 (Experimental): Randomized 3:1 for single ascending dose
  Interventions: Drug: REGN17092; Drug: Matching Placebo
- Expansion Cohort 3 (Experimental): Randomized 3:1 for single ascending dose
  Interventions: Drug: REGN17092; Drug: Matching Placebo

INTERVENTIONS:
Drug: REGN17092 — Single ascending intravenous (IV) or subcutaneous (SC) administration per the protocol
Drug: Matching Placebo — Single ascending IV or SC administration per the protocol

SUMMARY:
The purpose of this study is to learn about the safety and tolerability of different doses of REGN17092 administered with a needle either under the skin (called "subcutaneous") or into a vein (called an "infusion") in healthy participants. This is the first time that REGN17092 will be given to people.

Other aims are to assess:

* How much of the study drug is in the blood at different times
* Whether the body makes its own antibodies against the study drug (which could make the drug less effective or lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Has a SARS-CoV-2 negative test result from a sample collected ≤72 hours prior to randomization as described in the protocol
2. Has received complete primary series of standard-of-care COVID-19 vaccination per local guidance, completed at least 2 weeks prior to screening
3. Has a body mass index (BMI) between 18 and 31 Kg/m^2 (inclusive) at the screening visit
4. Is judged by the investigator to be in good health based on medical history, physical examination, vital sign measurements, and electrocardiogram (ECG)s performed at screening and/or prior to administration of initial dose of study drug

Key Exclusion Criteria:

1. History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, infectious, autoimmune, oncologic, psychiatric or neurological disease, as assessed by the investigator as described in the protocol
2. Presents any concern to the investigator that might confound the results of the study or poses an additional risk to the participant by their participation in the study
3. Was hospitalized (ie, >24 hours) for any reason within 30 days of the screening visit
4. Has history of alcohol or drug abuse as determined by the investigator
5. Has a history of significant multiple and/or severe allergies (eg, latex gloves), or has had an anaphylactic reaction to prescription or non-prescription drugs or food

NOTE: Other protocol defined inclusion / exclusion criteria apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of all treatment emergent adverse events (TEAEs) | Through approximately day 365
Severity of all TEAEs | Through approximately day 365
Occurrence of all treatment emergent serious adverse events (TE-SAEs) | Through approximately day 365
Severity of all TE-SAEs | Through approximately day 365

SECONDARY OUTCOMES:
Concentrations of REGN17092 in serum over time | Through approximately day 365
Incidence of Anti-drug antibodies (ADAs) to REGN17092 over time | Through approximately day 365
Titer of ADAs to REGN17092 over time | Through approximately day 365

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- UZ Leuven Gasthuisberg Campus, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

DOCUMENTS (1):
  • Informed Consent Form (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT05923424/ICF_000.pdf